CLINICAL TRIAL: NCT03161366
Title: An Open-label, Single Arm Study to Provide Additional Information on Safety and Effectiveness of rVSVΔG-ZEBOV-GP
Brief Title: Providing Additional Information on the Safety and Effectiveness of an Ebola Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Epicentre (Other)
Collaborators: Medecins Sans Frontieres, Netherlands (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V920-01
Record Dates: First submitted 2017-05-18; First posted 2017-05-19 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Ebola Virus Disease
Keywords: Ebola Zaire Outbreak; Safety of rVSVΔG-ZEBOV-GP vaccine; Effectiveness of rVSVΔG-ZEBOV-GP vaccine
MeSH Terms: conditions — Hemorrhagic Fever, Ebola

STUDY DESIGN:
Intervention Model Description: Interventional, single arm, open-label, non-randomized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): Vaccination of contacts and contacts of contacts of a confirmed Ebola Zaire case with one dose of rVSVΔG-ZEBOV-GP (≥ 2x10^7 PFU)
  Interventions: Biological: rVSVΔG-ZEBOV-GP

INTERVENTIONS:
Biological: rVSVΔG-ZEBOV-GP — Ring vaccination with vaccination of contacts and contacts of contacts after laboratory confirmation of one Ebola Zaire case

SUMMARY:
Interventional, single arm, open-label, non-randomized, phase IIIb study to accumulate additional data on safety and effectiveness of one dose of rVSVΔG-ZEBOV-GP against Ebola virus disease.

DETAILED DESCRIPTION:
Ebola Virus Disease remains ill-known by populations, creating fear and mistrust, is highly contagious, requiring strict isolation measures and with only supportive therapy available that has limited impact on case-fatality which remains high (30 -80%).1 Among vaccines in development, the rVSVΔG-ZEBOV-GP vaccine has given the most promising results in terms of efficacy and safety having been evaluated now in more than 10,000 individuals.

Ring vaccination is a known strategy to control epidemics with specific transmission chains and has been successfully implemented to eradicate smallpox. Ring vaccination enhances standard public health measures of contact tracing, isolation, and community engagement and could be effective when such measures are in place. Building on the interim results of the Ebola ça Suffit trial, there is a need for continued access to a vaccine of which available results suggest that it is safe and likely efficacious against EVD. Although only isolated cases have been reported in Guinea, Sierra Leone and Liberia in 2016, 10 the risk of resurgence or of continued isolated cases in West Africa remains. Moreover, a new outbreak with Ebola Zaïre could start any moment in any of the countries where previous outbreaks occurred as in for example Democratic Republic of Congo and Uganda.

However, the unusual design of the ring trial and the decision to abandon the control group because of strong evidence that the vaccine prevented disease means there may not be enough data to ensure approval from regulatory agencies. Therefore, additional information is still required to consolidate knowledge on the rVSVΔG-ZEBOV-GP vaccine to support regulatory approval and licensure for future access. Additional information is also needed on ring vaccination and contextual adaptations to this approach to ensure its feasibility and effectiveness in the control of Ebola outbreaks in potentially diverse contexts.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 6 years or older will be enrolled in the study if they are a contact or contact of contact of a laboratory-confirmed Ebola virus disease case. Children aged between 1 and 6 years may also be enrolled in the study in case there is a confirmed contact with a laboratory-confirmed Ebola patient
* willing to accept weekly visits
* intending to remain in the study area for three months
* providing informed consent, and where applicable, assent

Exclusion Criteria:

* history of EVD (self-report or laboratory confirmed)
* history of having received other investigational research agents in the previous 28 days
* history of anaphylaxis to a vaccine or vaccine component (self-report)
* severe illness that makes the person bed-bound or requiring hospitalization at the time of the vaccination
* severe immunocompromised status
* history of having received immunosuppressant therapies that would substantially interfere with the mode of action of the Ebola vaccine in the previous 6 months
* unwilling to accept weekly visits
* not intending to remain in the study area for three months
* informed consent or assent not provided
* any other condition in which, in the judgment of the investigator, would interfere with or serve as a contraindication to protocol adherence, or impair the subject or caregiver's ability to give informed consent, and where applicable, assent.
* fever above 38°C
* previous receipt of rVSVΔG-ZEBOV-GP in the last 3 years or at being part of another Ebola vaccine clinical trial.

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2018-05-28 (Actual); Primary Completion 2018-07-14 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Cumulative incidence | 84 days after vaccination
  Occurrence of Ebola Zaire cases amongst contacts and contacts of contacts

SECONDARY OUTCOMES:
Assessment of Adverse and Serious Adverse Events | 84 days after vaccination
  Safety of a single dose of rVSVΔG-ZEBOV-GP

CONTACTS AND LOCATIONS:
Locations (2):
- Médecins Sans Frontières, Kinshasa, Democratic Republic of the Congo
- Epicentre, Mbarara, Uganda

IPD SHARING:
Plan to Share IPD: Undecided
To be done following MSFdata sharing policy